CLINICAL TRIAL: NCT00522795
Title: BrUOG-E-215-Neoadjuvant Paclitaxel Poliglumex (PPX; CT-2103), Cisplatin and Radiation for Esophageal Cancer: A Phase II Trial. (CTI#X64001
Brief Title: Neoadjuvant Paclitaxel Poliglumex, Cisplatin and Radiation for Esophageal Cancer: A Phase II Trial (CTI#X64001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of Maryland Greenebaum Cancer Center (Other)
Responsible Party: Principal Investigator, howard safran, Principle Investigator, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-E-215
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — protein phosphatase 4; Cisplatin; Radiation; paclitaxel poliglumex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PPX with cisplatin and radiation (Experimental): PPX 50mg/m2 wk and cisplatin 25mg/m2 wk for 6 weeks with 50.4 GY concurrent radiation
  Interventions: Drug: PPX with cisplatin and radiation

INTERVENTIONS:
Drug: PPX with cisplatin and radiation — weekly IV treatment of Paclitaxel Poliglumex and Cisplatin for 6 weeks
  Other Names: Paclitaxel Poliglumex, Cisplatin and radiation

SUMMARY:
Neoadjuvant Paclitaxel Poliglumex (PPX; CT-2103), Cisplatin and Radiation for Esophageal Cancer: A Phase II Trial. (CTI#X64001

DETAILED DESCRIPTION:
32 patients with esophageal or gastroesophageal junction cancer will receive Radiation:50.4 Gy at 180cGy fraction/day for 28 treatments and Paclitaxel Poliglumex (PPX) and Cisplatin weekly times 6 followed by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients are required to have pathologically confirmed adenocarcinoma or squamous cell carcinoma of the esophagus or gastroesophageal junction
* Patients may have celiac adenopathy
* There must be no evidence of distant organ metastases
* No prior chemotherapy or radiation for esophageal cancer
* Patients must be > 18 years of age, and non pregnant
* Patients must have an ANC > 1,500/ul, platelets > 100,000/ul, creatinine < 2.0 and bilirubin < 1.5 x ULN-ECOG performance status 0-1.
* Female patients, must either be not of child bearing potential or have a negative pregnancy test within 14 days of starting study treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal. Pregnant or lactating females are not eligible
* No contraindications to esophagectomy
* Signed informed consent

Exclusion Criteria:

* Active or uncontrolled infection
* Patients must not have other coexistent medical condition that would preclude protocol therapy.
* Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-08; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Brown University
Locations (1):
- Lifespan Hospitals, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual closed in August 2009, 40 patients were enrolled
Groups:
- PPX, Cisplatin, Radiation: * PPX: 50 mg/m2/week days 1, 8, 15, 22, 29, 36.
  * Cisplatin: 25 mg/m2/week days 1, 8, 15, 22, 29, 36. Cisplatin, will be administered over ½ hour in 250 cc ns weekly for 6 weeks. Cisplatin will be administered after PPX
Period: Overall Study
Arm/Group | PPX, Cisplatin, Radiation
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PPX, Cisplatin, Radiation
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathologic Response
Description: Per pathology review post surgery
Time Frame: At Surgery approximately 4weeks after last treatment
Population: Twelve of 37 patients (32%) had pathologic complete responses. The 12 patients with pathologic CR all had adenocarcinoma.
Measure: Number; unit: participants
Arm/Group | PPX, Cisplatin, Radiation
Number analyzed (Participants) | 40
participants | 12

ADVERSE EVENTS:
Arm/Group | PPX, Cisplatin, Radiation
Serious Adverse Events (participants affected / at risk) | 14/40
Other Adverse Events (participants affected / at risk) | 2/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PPX, Cisplatin, Radiation (N=40)
esophagitis, nauseam dehydration, electrolyte imbalance, potassium and mood alteration (Investigations) | 1 (1)
allergic reaction/hypersensitivity (Investigations) | 1 (1)
nausea, dehydration, esophagitis, death (Investigations) | 1 (1) — death related to progressive disease and carcinoma meningitis
multiorgan failure (Investigations) | 1 (1) — post op esophagectomy 2 1/2 months post chemotherapy not related to chemotherapy
leukopenia, esophagitis, dehydration, nausea, vomiting, neutropenia, hypotension (Investigations) | 1 (1)
hyperglycemia, dehydration (Investigations) | 1 (1)
infection of gallbladder with normal ANC (Investigations) | 1 (1)
dysphagia, dizziness, dehydration (Investigations) | 1 (1)
hypokalemia, hypomagnesemia, weakness, anorexia, opportunistic infection (Investigations) | 1 (1)
thrombosis, hematoma, hypomagnesemia, extrapyramidal/restless (Investigations) | 1 (2)
nausea, vomiting, weakness, ischemic colitis (Investigations) | 1 (1)
thrombosis/embolism (Investigations) | 1 (1)
infection with normal ANC (cellulitis) and albumin (Investigations) | 1 (1)
pneumothorax (Investigations) | 1 (1)
DVT (Investigations) | 1 (1)
acute vascular leak, GI other, hypotension, anorexia, hypothermia,INR (Investigations) | 1 (1) — GI other is abdominal compartment syndrome
abdominal pain and dehydration (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PPX, Cisplatin, Radiation (N=40)
esophagitis (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No